CLINICAL TRIAL: NCT07028372
Title: Long Term Follow-up of Cardiac Arrest Survivors Exposed to Ultra-rapid Cooling, a Prospective Non-interventional Cohort
Brief Title: Long Term Follow-up of Cardiac Arrest Survivors Exposed to Ultra-rapid Cooling
Acronym: AFTERCOOL
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ORIXHA (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP250360; 2025-A00442-47 (Other: IDRCB number)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest (CA); Resuscitated Sudden Cardiac Death; Post Cardiac Arrest Patient Who Was Treated by Hypothermia Protocol
Keywords: Cardiac arrest; Hypothermia; Target temperature management; Liquid ventilation; Resuscitation; long-term outcomes
MeSH Terms: conditions — Heart Arrest; Hypothermia | interventions — Activities of Daily Living; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resuscitated OverCool clinical investigation participants alive at 28 days after cardiac arrest: Patients who were resuscitated after cardiac arrest, treated with ultrarapid cooling as part of the OverCool clinical investigation and survived until the end of the investigation (28 days after cardiac arrest and subsequent Vent2Cool treatment).
  Interventions: Other: Short Form Health Survey (SF-36); Other: Modified Rankin Score (mRS); Other: Activity of Daily Living (ADL) questionnaire; Other: New York Heart Association (NYHA) Classification; Other: St George's Respiratory Questionnaire (SGRQ)

INTERVENTIONS:
Other: Short Form Health Survey (SF-36) — Heath-related quality-of-life is assessed using the SF-36 questionnaire, which is administered at the inclusion visite, then at month 6, year 1, year 2, year 3, year 4 and year 5, in the form of a telephone interview.
Other: Modified Rankin Score (mRS) — The degree of disability/dependence is evaluated using the mRS scale at the inclusion visite, then at month 6, year 1, year 2, year 3, year 4 and year 5, via telephone interview.
Other: Activity of Daily Living (ADL) questionnaire — Level of independence is evaluated using the ADL questionnaire, which is administered at the inclusion visite, then at month 6, year 1, year 2, year 3, year 4 and year 5, in the form of a telephone interview.
Other: New York Heart Association (NYHA) Classification — The extent of heart failure is assessed using the NYHA functional classification at the inclusion visite, then at month 6, year 1, year 2, year 3, year 4 and year 5, via telephone interview.
Other: St George's Respiratory Questionnaire (SGRQ) — Respiratory status is assessed using the SGRQ questionnaire at the inclusion visite, then at month 6, year 1, year 2, year 3, year 4 and year 5, via telephone interview.

SUMMARY:
Less than 10% of patients eliciting out-of-hospital cardiac arrest (OHCA) survive, although 30% can be resuscitated by Emergency services before admission in Intensive Care Units (ICU). The majority succumb to Post-Cardiac Arrest Syndrome (PCAS). PCAS is associated with high mortality (60-70%) and morbidity.

One proposed method of preventing the neurological and cardiac consequences of PCAS is to lower the body temperature to 33°C as quickly as possible. This approach is known as therapeutic hypothermia or Targeted Temperature Management (TTM). The Vent2Cool system, developed by Orixha, is a novel approach that enables the rapid induction of therapeutic hypothermia by using hypothermic Total Liquid Ventilation (TLV) to reach a protective temperature of 33°C within minutes.

The OverCool feasibility study, which started in April 2025, is designed to validate the clinical performance and safety of an ultra-rapid cooling approach combining ultra-rapid hypothermia induction using the Vent2Cool system, and maintenance and rewarming using the ArcticSun system.

The AfterCool study aims to evaluate long-term outcomes during a five-year follow-up of cardiac arrest survivors who were treated with ultrarapid cooling in the OverCool study.

DETAILED DESCRIPTION:
Fewer than 10% of patients experiencing out-of-hospital cardiac arrest (OHCA) survive, although 30% can be resuscitated by emergency services before being admitted to intensive care units (ICUs). Many cardiac arrest patients who are initially resuscitated by first responders and/or EMS, however, are condemned to a 'second death' in the ICU due to severe neurological and multi-visceral sequelae from post-cardiac arrest syndrome (PCAS).

One proposed method of preventing the neurological and cardiac complications of PCAS is to lower the body temperature to 33°C as quickly as possible. This approach is known as therapeutic hypothermia or Targeted Temperature Management (TTM). However, the cooling power of available technologies is insufficient to induce therapeutic hypothermia, and they do not improve outcomes for most patients. Conversely, experimental reports clearly demonstrate that therapeutic hypothermia can dramatically improve clinical outcomes if applied within two to three hours of resuscitation.

The devices currently available for TTM are mostly external cooling devices, such as blankets, pads and suits. These devices have a cooling performance of less than 1°C per hour in the body's core and in vital organs with high blood flow. Orixha's Vent2Cool is a novel approach that enables the induction of ultra-rapid therapeutic hypothermia (URTH) by using hypothermic total liquid ventilation (TLV) to reach a protective temperature of 33°C within minutes.

The OverCool feasibility study, which has been approved by the French authorities and began enrolment in early 2025, is designed to test the feasibility of ultra-rapid cooling. It aims to validate the clinical performance and safety of an ultra-rapid cooling approach combining ultra-rapid hypothermia induction using the Vent2Cool system, and maintenance and rewarming using the ArcticSun system. OverCool will pave the way for other clinical investigations to demonstrate the superior clinical benefits of this new approach to hypothermic TTM compared to the standard of care.

The AfterCool study will follow cardiac arrest survivors who were treated with ultrarapid cooling in the Overcool study for five years. The AfterCool approach aligns with the need to evaluate long-term outcomes after cardiac arrest, as endorsed by the French AfterROSC network, which supports research into post-cardiac arrest patients.

Eligible subjects, after having received clear, impartial and complete information, and not having objected to participation in the study, will be included. At the inclusion visit, a detailed questionnaire regarding life status, quality of life, putative rehospitalization, cardiovascular, neurological and respiratory status will be administered.

At 6±1 months and 12±1 months after inclusion, and then yearly during a total period of 5 years, the patients or trusted persons or the close relatives or parents will be interviewed by phone, using the same questionnaire regarding life status, quality of life, putative rehospitalization, cardiovascular, neurological and respiratory status.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and over
* Cardiac arrest patient included in and alive at the end of the OverCool clinical investigation (28 days after the cardiac arrest)
* Non-opposition from the patient or the trusted person or the close relative or parent obtained within 3 months after the end of the OverCool study

Exclusion Criteria:

* Follow-up refusal from patient of trusted person or the close relative or parent
* Having being included in the OverCool clinical investigation but not submitted to the Vent2Cool procedure
* Impossibility to reach the patient or the trusted person or the close relative or parent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest patient included in and alive at the end of the OverCool clinical investigation (28 days after the cardiac arrest)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Life status at 5 years | 5 years
  The primary endpoint is the life status at 5 years assessed by phone interview. Whenever possible, life status will be confirmed by reviewing the medical record.

SECONDARY OUTCOMES:
Suspected cause of death | 5 years
  The suspected cause of death in the event of a death. Data are collected via interview. If the deceased is rehospitalised or receives additional care in a hospital that shares a medical database with centres participating in the Aftercool study, the information will be confirmed by reviewing the medical record.
Rehospitalization | 5 years
  Data are collected via interview. If a participant is rehospitalised or requires additional hospital care, and if that hospital shares a medical database with the centres of the Aftercool study, the information will be confirmed by reviewing the medical record.
Modified Rankin Scale (mRS) Score | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  The mRS scale is used to assess neurological status. mRS scale ranges from 0 (no residual symptoms) to 6 (dead). Higher scores indicate greater disability.
36-Item Short Form Health Survey (SF-36) score | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  The SF-36 questionnaire is a health-related quality of life scale, comprising eight scaled scores: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. Scores range from 0 - 100. Higher scores mean less disability.
Activity of Daily Living (ADL) score | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  Autonomy level is measured using a six-item ADL scale. Scores range from 0 (the patient is very dependent) to 6 (the patient is independent).
Cardiovascular adverse events | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  Cardiovascular adverse events that occurred between interviews: acute coronary syndromes, arrhythmias, stroke or other cerebrovascular events.
NewYork Health Association (NYHA) status | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  The extent of heart failure is assessed using The New York Heart Association (NYHA) Functional Classification. It enables patients to be classified into classes I to IV according to their symptoms, with class I corresponding to the best health.
Respiratory adverse events | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  Respiratory adverse events that occurred between interviews.
St-George's Respiratory Questionnaire (SGRQ) Score | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  The SGRQ questionnaire (PDF) has 50 items divided into three parts measuring symptoms, activity limitation and social and emotional impact of disease. Scores range from 0 to 100, with higher scores indicating more limitations
Home oxygen therapy | Baseline, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  The need to resort to the use of home oxygen therapy between interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Alain CARIOU, MD PhD, Principal Investigator — AP-HP, Cochin Hospital, Intensive Care and Resuscitation Department
Locations (2):
- France (2):
  - Angers University Hospital, Medical Intensive Care Unit, Vent'Lab, Angers
  - AP-HP Centre, Cochin Hospital, Medical Intensive Care Unit, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tissier R, Taccone FS, Lamhaut L, Vicaut E, Paublant F, Ricard JD, Mercat A, Cariou A. Design of the OverCool study: Lung-conservative liquid ventilation for the induction of Ultra-Rapid Cooling after Cardiac Arrest (OverCool). Resusc Plus. 2025 Mar 10;23:100926. doi: 10.1016/j.resplu.2025.100926. eCollection 2025 May. PMID 40212905
- [Background] Dumas F, Paoli A, Paul M, Savary G, Jaubert P, Chocron R, Varenne O, Mira JP, Charpentier J, Bougouin W, Cariou A. Association between previous health condition and outcome after cardiac arrest. Resuscitation. 2021 Oct;167:267-273. doi: 10.1016/j.resuscitation.2021.06.017. Epub 2021 Jul 7. PMID 34245838
- [Background] Bougouin W, Lascarrou JB, Chelly J, Benghanem S, Geri G, Maizel J, Fage N, Sboui G, Pichon N, Daubin C, Sauneuf B, Mongardon N, Taccone F, Hermann B, Colin G, Lesieur O, Deye N, Chudeau N, Cour M, Bourenne J, Klouche K, Klein T, Raphalen JH, Muller G, Galbois A, Bruel C, Jacquier S, Paul M, Sandroni C, Cariou A. Performance of the ERC/ESICM-recommendations for neuroprognostication after cardiac arrest: Insights from a prospective multicenter cohort. Resuscitation. 2024 Sep;202:110362. doi: 10.1016/j.resuscitation.2024.110362. Epub 2024 Aug 14. PMID 39151721
- [Background] Flajoliet N, Bourenne J, Marin N, Chelly J, Lascarrou JB, Daubin C, Bougouin W, Cariou A, Geri G. Return to work after out of hospital cardiac arrest, insights from a prospective multicentric French cohort. Resuscitation. 2024 Jun;199:110225. doi: 10.1016/j.resuscitation.2024.110225. Epub 2024 Apr 27. PMID 38685375
- [Background] Lascarrou JB, Merdji H, Le Gouge A, Colin G, Grillet G, Girardie P, Coupez E, Dequin PF, Cariou A, Boulain T, Brule N, Frat JP, Asfar P, Pichon N, Landais M, Plantefeve G, Quenot JP, Chakarian JC, Sirodot M, Legriel S, Letheulle J, Thevenin D, Desachy A, Delahaye A, Botoc V, Vimeux S, Martino F, Giraudeau B, Reignier J; CRICS-TRIGGERSEP Group. Targeted Temperature Management for Cardiac Arrest with Nonshockable Rhythm. N Engl J Med. 2019 Dec 12;381(24):2327-2337. doi: 10.1056/NEJMoa1906661. Epub 2019 Oct 2. PMID 31577396
- [Background] Arrich J, Herkner H, Mullner D, Behringer W. Targeted temperature management after cardiac arrest. A systematic review and meta-analysis of animal studies. Resuscitation. 2021 May;162:47-55. doi: 10.1016/j.resuscitation.2021.02.002. Epub 2021 Feb 12. PMID 33582259
- [Background] Kohlhauer M, Lidouren F, Remy-Jouet I, Mongardon N, Adam C, Bruneval P, Hocini H, Levy Y, Blengio F, Carli P, Vivien B, Ricard JD, Micheau P, Walti H, Nadeau M, Robert R, Richard V, Mulder P, Maresca D, Demene C, Pernot M, Tanter M, Ghaleh B, Berdeaux A, Tissier R. Hypothermic Total Liquid Ventilation Is Highly Protective Through Cerebral Hemodynamic Preservation and Sepsis-Like Mitigation After Asphyxial Cardiac Arrest. Crit Care Med. 2015 Oct;43(10):e420-30. doi: 10.1097/CCM.0000000000001160. PMID 26110489
- [Background] Darbera L, Chenoune M, Lidouren F, Kohlhauer M, Adam C, Bruneval P, Ghaleh B, Dubois-Rande JL, Carli P, Vivien B, Ricard JD, Berdeaux A, Tissier R. Hypothermic liquid ventilation prevents early hemodynamic dysfunction and cardiovascular mortality after coronary artery occlusion complicated by cardiac arrest in rabbits. Crit Care Med. 2013 Dec;41(12):e457-65. doi: 10.1097/CCM.0b013e3182a63b5d. PMID 24126441
- [Background] Che D, Li L, Kopil CM, Liu Z, Guo W, Neumar RW. Impact of therapeutic hypothermia onset and duration on survival, neurologic function, and neurodegeneration after cardiac arrest. Crit Care Med. 2011 Jun;39(6):1423-30. doi: 10.1097/CCM.0b013e318212020a. PMID 21610611
- [Background] Dankiewicz J, Cronberg T, Lilja G, Jakobsen JC, Levin H, Ullen S, Rylander C, Wise MP, Oddo M, Cariou A, Belohlavek J, Hovdenes J, Saxena M, Kirkegaard H, Young PJ, Pelosi P, Storm C, Taccone FS, Joannidis M, Callaway C, Eastwood GM, Morgan MPG, Nordberg P, Erlinge D, Nichol AD, Chew MS, Hollenberg J, Thomas M, Bewley J, Sweet K, Grejs AM, Christensen S, Haenggi M, Levis A, Lundin A, During J, Schmidbauer S, Keeble TR, Karamasis GV, Schrag C, Faessler E, Smid O, Otahal M, Maggiorini M, Wendel Garcia PD, Jaubert P, Cole JM, Solar M, Borgquist O, Leithner C, Abed-Maillard S, Navarra L, Annborn M, Unden J, Brunetti I, Awad A, McGuigan P, Bjorkholt Olsen R, Cassina T, Vignon P, Langeland H, Lange T, Friberg H, Nielsen N; TTM2 Trial Investigators. Hypothermia versus Normothermia after Out-of-Hospital Cardiac Arrest. N Engl J Med. 2021 Jun 17;384(24):2283-2294. doi: 10.1056/NEJMoa2100591. PMID 34133859
- [Background] Sandroni C, Nolan JP, Andersen LW, Bottiger BW, Cariou A, Cronberg T, Friberg H, Genbrugge C, Lilja G, Morley PT, Nikolaou N, Olasveengen TM, Skrifvars MB, Taccone FS, Soar J. ERC-ESICM guidelines on temperature control after cardiac arrest in adults. Intensive Care Med. 2022 Mar;48(3):261-269. doi: 10.1007/s00134-022-06620-5. Epub 2022 Jan 28. PMID 35089409
- [Background] Boissady E, Kohlhauer M, Lidouren F, Hocini H, Lefebvre C, Chateau-Jouber S, Mongardon N, Deye N, Cariou A, Micheau P, Ghaleh B, Tissier R. Ultrafast Hypothermia Selectively Mitigates the Early Humoral Response After Cardiac Arrest. J Am Heart Assoc. 2020 Dec;9(23):e017413. doi: 10.1161/JAHA.120.017413. Epub 2020 Nov 17. PMID 33198571
- [Background] Kohlhauer M, Boissady E, Lidouren F, de Rochefort L, Nadeau M, Rambaud J, Hutin A, Dubuisson RM, Guillot G, Pey P, Bruneval P, Fortin-Pellerin E, Sage M, Walti H, Cariou A, Ricard JD, Berdeaux A, Mongardon N, Ghaleh B, Micheau P, Tissier R. A new paradigm for lung-conservative total liquid ventilation. EBioMedicine. 2020 Feb;52:102365. doi: 10.1016/j.ebiom.2019.08.026. Epub 2019 Aug 22. PMID 31447395
- [Background] Chenoune M, Lidouren F, Adam C, Pons S, Darbera L, Bruneval P, Ghaleh B, Zini R, Dubois-Rande JL, Carli P, Vivien B, Ricard JD, Berdeaux A, Tissier R. Ultrafast and whole-body cooling with total liquid ventilation induces favorable neurological and cardiac outcomes after cardiac arrest in rabbits. Circulation. 2011 Aug 23;124(8):901-11, 1-7. doi: 10.1161/CIRCULATIONAHA.111.039388. Epub 2011 Aug 1. PMID 21810660
- [Background] Berdowski J, Berg RA, Tijssen JG, Koster RW. Global incidences of out-of-hospital cardiac arrest and survival rates: Systematic review of 67 prospective studies. Resuscitation. 2010 Nov;81(11):1479-87. doi: 10.1016/j.resuscitation.2010.08.006. Epub 2010 Sep 9. PMID 20828914
- [Background] Lemiale V, Dumas F, Mongardon N, Giovanetti O, Charpentier J, Chiche JD, Carli P, Mira JP, Nolan J, Cariou A. Intensive care unit mortality after cardiac arrest: the relative contribution of shock and brain injury in a large cohort. Intensive Care Med. 2013 Nov;39(11):1972-80. doi: 10.1007/s00134-013-3043-4. Epub 2013 Aug 14. PMID 23942856
- [Background] Dumas F, Bougouin W, Perier MC, Marin N, Goulenok C, Vieillard-Baron A, Diehl JL, Legriel S, Deye N, Cronier P, Ricome S, Chemouni F, Mekontso Dessap A, Beganton F, Marijon E, Jouven X, Empana JP, Cariou A. Long-term follow-up of cardiac arrest survivors: Protocol of the DESAC (Devenir des survivants d'Arrets Cardiaques) study, a French multicentric prospective cohort. Resusc Plus. 2023 Aug 31;16:100460. doi: 10.1016/j.resplu.2023.100460. eCollection 2023 Dec. PMID 37693335